CLINICAL TRIAL: NCT00828594
Title: A Phase 1 Open Label/ Phase 2 Randomized, Double-blind, Multicenter Study Investigating the Combination of RAD001 and Sorafenib (Nexavar®) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Global Study Looking at the Combination of RAD001 and Sorafenib to Treat Patients With Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001O2101
Record Dates: First submitted 2009-01-09; First posted 2009-01-26 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; dose-finding study; randomized trial; medical treatment; RAD001; sorafenib; Advanced hepatocellular cancer (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Everolimus; Sorafenib

ARMS (1):
- Phase 1: RAD001 plus sorafenib (Experimental)
  Interventions: Drug: RAD001; Drug: RAD001, sorafenib

INTERVENTIONS:
Drug: RAD001
Drug: RAD001, sorafenib

SUMMARY:
Phase 1 Evaluate the safety and tolerability of RAD001 in combination with sorafenib in patients with advance hepatocellular cancer (HCC) and to determine the maximum tolerated dose (MTD)

Phase 2 To estimate the treatment effect as a measure of anti-tumor activity in terms of Time to Progression (TTP) of the combination of RAD001 plus sorafenib, at the MTD, as compared to sorafenib alone

ELIGIBILITY:
Inclusion Criteria:

* Advanced liver cancer
* No previous systemic therapy for liver cancer
* Measurable disease on CT or MRI
* ECOG 1 or less
* Child-Pugh A

Exclusion Criteria:

* Active bleeding during the last 30 days
* Known history of HIV seropositivity
* Any severe and/or uncontrolled medical conditions including

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of combination RAD001+sorafenib | Until maximum tolerated dose is determined
Time to disease progression assessed when 60 events have been observed | Until number of events are reached

SECONDARY OUTCOMES:
Safety and tolerability of the combination of RAD001 plus sorafenib as measured by the rate and severity of adverse events | Estimate of 1 year for each patient - Until all patients have disease progression or leave study due to intolerable toxicity
Tumor response | Estimate of 1 year for each patient - Until all patients have disease progression or leave study due to intolerable toxicity
Biomarkers- effect of treatment on soluble markers of angiogenesis and apoptosis | Estimate of 1 year for each patient - Until all patients have disease progression or leave study due to intolerable toxicity
Overall tumor response (phase 2) | Estimate of 1 year for each patient - Until number of events reached and final analysis
Progression Free Survivor, Overall Survivor (phase 2) | Estimate of 1 year for each patient - Until number of events reached and final analysis
Safety and tolerability - of the combination of RAD001 plus sorafenib as measured by the rate and severity of adverse events (phase 2) | Estimate of 1 year for each patient - Until number of events reached and final analysis
Pharmokinetics of RAD001 at pre-dose and 1 hour and 2 hours post-dose (phase 2) | Estimate of 1 year for each patient - Until number of events reached and final analysis
Biomarkers effect of treatment on soluble markers of angiogenesis and apoptosis (phase 2) | Estimate of 1 year for each patient - Until number of events reached and final analysis
Pharmokinetics of RAD001 at pre-dose and 1 hour and 2 hours post-dose | Estimate of 1 year for each patient - Until all patients have disease progression or leave study due to intolerable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - UCLA Department of Medicine, Los Angeles, California
  - Duke University, Durham, North Carolina
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Invstigative Site, Madrid
- Novartis Investigative Site, Tainan, Taiwan